CLINICAL TRIAL: NCT05780593
Title: Effects of Manual Therapy and Inclined Board Standing on Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agile Institute of Rehabilitation Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AgileRehab
Record Dates: First submitted 2023-03-13; First posted 2023-03-22 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Manual Therapy; Passive Stretching; Inclined Board Standing
MeSH Terms: conditions — Low Back Pain | interventions — Musculoskeletal Manipulations; Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Two arm parallel research involves two groups randomized into Interventional Group-A and Interventional Group-B. The unit of randomization will be Agile Institute of Rehabilitation Sciences. This study will use 2 (between groups: Effects of mobilization with passive stretching of lateral rotators along with inclined board standing vs Inclined board standing) ×3 (time: before vs. after vs. 4 weeks after follow-up) mixed design to measure the effects of mobilization, passive stretching of hip abductors and inclined board standing on low back patient.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group A (Experimental): Manual mobilization of lumbosacral spine along with passive stretching of the hip abductors and 01 minute of inclined board standing for 03 times a day.
  Interventions: Other: Manual Therapy; Other: Inclined Board Standing
- Intervention Group B (Experimental): Routine medications(if any) along with 01 minute of inclined board standing for 03 times a day.
  Interventions: Other: Inclined Board Standing

INTERVENTIONS:
Other: Manual Therapy — After the baseline assessment, each intervention group will be given physical therapy treatment. The group A will receive Manual Mobilization of the Lumbosacral Spine followed by passive stretching of the hip abductors of both sides of the body. The patient then will be asked to stand on the inclined board for 01 minute with feet 3 to 4 inches apart hands placed on the wall at the level of shoulder joints. After 01-minute patient will be asked to leave the inclined board. The patient will be advised to do this 01-minute inclined board standing for three times a day at home. All the patients in Group A will receive this treatment regime for two weeks.
  Other Names: Passive Stretching; Inclined Board Standing
  Arms: Intervention Group A
Other: Inclined Board Standing — The patients in Group B will be asked to stick to their medications if advised and stand on the inclined board for 01 minute. Inclined boards will be provided to all patients and will be advised to follow the inclined standing for 01 minute for three times a day at home for two weeks. After two weeks at the completion of intervention, they will be assessed through self-reporting questionnaires of the study.
  Other Names: Routine medications(if any)

SUMMARY:
To date, there have been limited clinical trials conducted to determine the effects of manual therapy combined with passive stretching and inclined board standing for treating low-back pain. This will be the first randomized controlled trial to evaluate the effects of these integrated interventions. The study aims to develop a new approach towards the cost-effective management of low-back pain, in line with the World Health Organization's (WHO) vision of maximizing health outcomes, preventing disability, and reducing the cost of care.

DETAILED DESCRIPTION:
Manual therapy is a sub-type of physical therapy that uses hands-on maneuver to diagnose and treat musculoskeletal pain and dysfunction. Mobilization and manipulation are widely used for the management of low-back-pain (LBP), a common and debilitating condition that affects millions of people worldwide. The goal of manual therapy is to improve mobility, reduce pain and discomfort, and enhance functional capacity. Evidence is growing now a days that is in the direction of usage of manual therapy for the treatment of the lower back pain. Many studies have demonstrated the effectiveness of manual-therapy procedures such as spinal high velocity low amplitude thrust, low velocity and high intensity joint passive movement, and massage in alleviating pain and dysfunction and enhancing physical and mental functions in clinical cases with lower backache.

The prime purpose of this research aimed to investigate the relationship between the length of the tensor fasciae lata (TFL) and pelvic rotation during one-leg stance in healthy adults. 41 participants were assessed using a 3-dimensional motion analyzer, and their TFL length and hip rotation range of motion were measured. The results divided participants into two groups based on their pelvic rotation during one-leg stance. Although there was no significant difference in TFL length between the two groups, the study suggests that pelvic instability may cause trunk instability during one-leg stance.

Another study looked at static balance in three different standing positions with and without a foam surface. It found that standing over slanted surfaces increased postural unsteadiness, and that dorsiflexed ankles over a foam surface created more postural instability.

To create a human-like biped posture, a study created a Neural Controllable (NC) model to represent a human-like biped posture. The model generated physiologically reasonable muscle activations and captured the idea that individuals choose a low active stiffness level while standing to use less energy.

Another researcher reviewed the involvement of the "kinetic chain" in overhead athletes and applied it to clinical workout adjustments for the prevention and treatment of shoulder injuries. The study found that lower extremities, trunk, and scapular area all play a role in the formation of adequate terminal segment acceleration during overhead throwing and serving actions. The study suggests that traditional shoulder exercises should include scapular stabilizer and core musculature activation in addition to rotator cuff activation.

Research Gap:

Low-back-pain (LBP) is a Musculo-skeletal ailment that has a negative societal impact and is extremely common around the world, causing disability. LBP is one of the most common reasons people seek medical attention in the United States, along with neck pain, which is connected with the greatest healthcare expenses. Surgical patients are the most expensive per care episode, however the vast majority of lower backache management spending can be attributable to the substantially higher number of non-operative care episodes.

In 2021, Academy of Orthopedic Physical Therapy (AOPT) has published updated Clinical Practice Guidelines (CPG) for acute and chronic low-back-pain linked to the ICF model for physical therapists The updated Clinical Practice Guidelines (CPGs) for the treatment of lower back pain (LBP) recommend four interventional categories: exercise, manual and other-directed therapies, classification systems, and patient education. The guidelines were developed to be applicable globally and acknowledge that differences in factors such as healthcare systems, cultural norms, and social health determinants may impact the implementation of these recommendations. Physical therapists are the primary audience, but other stakeholders may also find the guidelines useful. The CPG update has identified knowledge gaps in the treatment of LBP and recommended further research using Single Level I RCT or Small-Sample Level II RCTs With Short Follow-up Times to develop better and cost-effective management approaches.

ELIGIBILITY:
Inclusion Criteria:

Participants are capable of receiving the treatment thrice a week willingly for maximum of 60 minutes.

Persistent low back pain that has lasted more than three months with no evidence of improvement, with or without discomfort into the lower limbs.

Low back pain on Numerical Pain Rating scale of at least 2/10 and less or equal to 9/10. Age 18-65 years

Exclusion Criteria:

No informed consent Pregnancy reported by the patient Prior surgical history of spine Previously diagnosed inflammatory joint disease. Warning complaints diagnosed by therapist. These cases were referred for lab investigation.

Motor or sensory neurological signs Cases of low-back-pain are not compliant with the exercise program. Previously or currently indulge in the exercise plan or physical fitness plan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
NEUMERIC PAIN RATING SCALE (NPRS) | 03 Months
  Changes from baseline numeric pain rating scale is a scale for pain starting from 0-10.

SECONDARY OUTCOMES:
Oswestry-Disability-Index (ODI) | 03 Months
  The ODI was established in English and has now been translated into over 40 languages. It was developed to measure the low back pain and disability over time. It consists of 10, with five-part sections. At the last, score is calculated by dividing the obtained score by total (50) multiplied by 100.
Short-form-12 questionnaire (SF-12) | 03 Months
  The Medical Outcomes Study (MOS), a multi-year study of patients with chronic illnesses, developed the 12-item Short Form Health Survey (SF-12). The SF-12 is a general HRQoL assessment that assesses general health status in eight dimensions (physical functioning, role limitations due to physical problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health).

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hafeez, Principal Investigator — Agile Institute of Rehabilitation Sciences; Muhammad Hafeez, Study Chair — The Islamia University of Bahawalpur
Locations (1):
- Agile Institute of Rehabilitation Center, Chak Four Hundred Fifty-four, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams, M. A., Bogduk, N., Burton, K., & Dolan, P. (2012). The Biomechanics of Back Pain-E-Book: Elsevier health sciences.
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Background] Alwadani FA, Liang H, Aruin AS. Effects of Ankle Angular Position and Standing Surface on Postural Control of Upright Stance. Motor Control. 2020 Jan 23;24(2):291-303. doi: 10.1123/mc.2019-0079. PMID 31972537
- [Background] Azevedo, R., Johnson, A., & Burkett, C. (2015). Does Training of Cognitive and Metacognitive Regulatory Processes Enhance Learning and Deployment of Processes with Hypermedia? Paper presented at the CogSci.
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Bialosky JE, Beneciuk JM, Bishop MD, Coronado RA, Penza CW, Simon CB, George SZ. Unraveling the Mechanisms of Manual Therapy: Modeling an Approach. J Orthop Sports Phys Ther. 2018 Jan;48(1):8-18. doi: 10.2519/jospt.2018.7476. Epub 2017 Oct 15. PMID 29034802
- [Background] Bialosky JE, Bishop MD, Price DD, Robinson ME, George SZ. The mechanisms of manual therapy in the treatment of musculoskeletal pain: a comprehensive model. Man Ther. 2009 Oct;14(5):531-8. doi: 10.1016/j.math.2008.09.001. Epub 2008 Nov 21. PMID 19027342
- [Background] Bishop MD, Torres-Cueco R, Gay CW, Lluch-Girbes E, Beneciuk JM, Bialosky JE. What effect can manual therapy have on a patient's pain experience? Pain Manag. 2015;5(6):455-64. doi: 10.2217/pmt.15.39. Epub 2015 Sep 24. PMID 26401979
- [Background] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405
- [Background] Buchbinder R, van Tulder M, Oberg B, Costa LM, Woolf A, Schoene M, Croft P; Lancet Low Back Pain Series Working Group. Low back pain: a call for action. Lancet. 2018 Jun 9;391(10137):2384-2388. doi: 10.1016/S0140-6736(18)30488-4. Epub 2018 Mar 21. PMID 29573871
- [Background] Chiarotto A, Deyo RA, Terwee CB, Boers M, Buchbinder R, Corbin TP, Costa LO, Foster NE, Grotle M, Koes BW, Kovacs FM, Lin CW, Maher CG, Pearson AM, Peul WC, Schoene ML, Turk DC, van Tulder MW, Ostelo RW. Core outcome domains for clinical trials in non-specific low back pain. Eur Spine J. 2015 Jun;24(6):1127-42. doi: 10.1007/s00586-015-3892-3. Epub 2015 Apr 5. PMID 25841358
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Background] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424
- [Background] Haddad C, Sacre H, Obeid S, Salameh P, Hallit S. Validation of the Arabic version of the "12-item short-form health survey" (SF-12) in a sample of Lebanese adults. Arch Public Health. 2021 Apr 23;79(1):56. doi: 10.1186/s13690-021-00579-3. PMID 33892801
- [Background] Hall AM, Scurrey SR, Pike AE, Albury C, Richmond HL, Matthews J, Toomey E, Hayden JA, Etchegary H. Physician-reported barriers to using evidence-based recommendations for low back pain in clinical practice: a systematic review and synthesis of qualitative studies using the Theoretical Domains Framework. Implement Sci. 2019 May 7;14(1):49. doi: 10.1186/s13012-019-0884-4. PMID 31064375
- [Background] Hultman G, Saraste H, Ohlsen H. Anthropometry, spinal canal width, and flexibility of the spine and hamstring muscles in 45-55-year-old men with and without low back pain. J Spinal Disord. 1992 Sep;5(3):245-53. doi: 10.1097/00002517-199209000-00001. PMID 1387820
- [Background] Jenkinson C, Layte R, Jenkinson D, Lawrence K, Petersen S, Paice C, Stradling J. A shorter form health survey: can the SF-12 replicate results from the SF-36 in longitudinal studies? J Public Health Med. 1997 Jun;19(2):179-86. doi: 10.1093/oxfordjournals.pubmed.a024606. PMID 9243433
- [Background] Kim DH, Park JK, Jeong MK. Influences of posterior-located center of gravity on lumbar extension strength, balance, and lumbar lordosis in chronic low back pain. J Back Musculoskelet Rehabil. 2014;27(2):231-7. doi: 10.3233/BMR-130442. PMID 24284274
- [Background] Negrini S, Giovannoni S, Minozzi S, Barneschi G, Bonaiuti D, Bussotti A, D'Arienzo M, Di Lorenzo N, Mannoni A, Mattioli S, Modena V, Padua L, Serafini F, Violante FS. Diagnostic therapeutic flow-charts for low back pain patients: the Italian clinical guidelines. Eura Medicophys. 2006 Jun;42(2):151-70. No abstract available. PMID 16767064
- [Background] Vincent-Onabajo GO, Nweze E, Kachalla Gujba F, Ali Masta M, Usman Ali M, Alhaji Modu A, Umeonwuka C. Prevalence of Low Back Pain among Undergraduate Physiotherapy Students in Nigeria. Pain Res Treat. 2016;2016:1230384. doi: 10.1155/2016/1230384. Epub 2016 Feb 3. PMID 26955486